CLINICAL TRIAL: NCT04042389
Title: Influence of WhatsApp and Electronic Mail Reminders on Oral Hygiene Compliance of Orthodontic Patients Using Planimetry
Brief Title: Oral Hygiene Reminders in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahsa University (Other)
Responsible Party: Principal Investigator, Kirti Saxena, Lecturer, Mahsa University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RMC/EC23/2017
Record Dates: First submitted 2019-07-28; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Compliance, Treatment
Keywords: WhatsApp; Email; Oral hygiene; Compliance; Orthodontics; Planimetry; Reminders
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WhatsApp (Experimental): WhatsApp reminders
  Interventions: Behavioral: WhatsApp reminder
- Email (Experimental): Email reminders
  Interventions: Behavioral: Email reminder
- Control (Other): No reminder
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: WhatsApp reminder — The WhatsApp group received oral health messages once a week for four weeks (totaling 4 messages) as a reminder to practice good oral hygiene
  The reminder included an image reminding them to maintain their oral hygiene.
  Other Names: Reminders
  Arms: WhatsApp
Behavioral: Email reminder — The Email group received oral health messages once a week for four weeks (totaling 4 messages) as a reminder to practice good oral hygiene
  The reminder included an image reminding them to maintain their oral hygiene.
  Other Names: Reminder
  Arms: Email
Behavioral: Control — No messages sent.
  Arms: Control

SUMMARY:
Objective: To determine the effect of WhatsApp and Email reminders on oral hygiene compliance of orthodontic patients.

Methods: A Randomized, parallel group, double blinded study was conducted on 54 patients undergoing orthodontic treatment at MAHSA University. They were randomized to 3 groups, namely WhatsApp (W) group, Email (E) group and Control (C) group with 18 subjects in each group. Group (W) and Group (E) received oral health messages once a week through WhatsApp and E-mail reminders respectively, while Group (C) did not receive any reminders. Plaque was measured at baseline (T0), after 4 weeks (T1), and after 8 weeks (T2). For each subject, two intraoral photographs were taken after application of plaque disclosing agent; and the area covered by plaque was measured on 12, 13, 43, 22, 23 and 33 teeth by planimetry.

DETAILED DESCRIPTION:
Fifty-four patients undergoing orthodontic treatment were recruited from the dental clinic of MAHSA University between Jan 2018 to April 2018. Voluntary written informed consent was obtained from all the subjects before the start of the study. They were randomly assigned into 3 groups namely WhatsApp (W) group, Email (E) group and Control (C) group with 18 subjects in each group. Oral hygiene messages through WhatsApp and Email were sent once a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients having fixed maxillary and mandibular orthodontic appliances with 0.022 AO conventional metal brackets,
* Aged ≥ 15 years,
* Undergone 3 months of orthodontic treatment,
* No significant medical or dental history
* Have access to cellular telephone and are online daily

Exclusion Criteria:

* Patients undergoing single arch treatment
* Missing maxillary lateral incisor, maxillary canine and mandibular canine
* Patients' orthodontic treatment duration < 3 months and > 4 months.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-04-29 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Change in plaque from baseline to 4 weeks | baseline (T0) to end of 4 weeks (T1)
  Plaque disclosing solution was applied to the pre-selected teeth (12,13,43, 22, 23, 33) followed by measurement of plaque using planimetry. All photographs were taken using a Canon Electro-Optical System (EOS) 550D (camera specifications). Plaque was analyzed using Image J software. Change in plaque score is assessed from baseline to 4 weeks in all the three groups.
  In the photo, region of interest targeted by the study was manually outlined using "Polygon selection tool", the total pixel present in this region is calculated by tracing tool. The pixel of the plaque area is determined by adjusting the color threshold to desirable range of value. The plaque sore was calculated in the form of percent covering tooth structure and the value of plaque on each tooth was determined and mean plaque was calculated.
Change in plaque from baseline to 8 weeks | Baseline (T0) to end of 8 weeks (T2)
  Plaque disclosing solution was applied to the pre-selected teeth (12,13,43, 22, 23, 33) followed by measurement of plaque using planimetry. All photographs were taken using a Canon EOS 550D (camera specifications). Plaque was analyzed using Image J software. Change in plaque score is assessed from baseline to 8 weeks in all the three groups.
  In the photo, region of interest targeted by the study was manually outlined using "Polygon selection tool", the total pixel present in this region is calculated by tracing tool. The pixel of the plaque area is determined by adjusting the color threshold to desirable range of value. The plaque sore was calculated in the form of percent covering tooth structure and the value of plaque on each tooth was determined and mean plaque was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Kirti Saxena, MDS, Principal Investigator — Mahsa University
Locations (1):
- MAHSA UNivesity, Jenjarum, Selangor, Malaysia